CLINICAL TRIAL: NCT06231901
Title: Comparison of Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach and Goal-Directed Training on Occupational Performance and Functional Status in Children With Cerebral Palsy: A Three-Armed Randomized Controlled Trial
Brief Title: Comparison of CO-OP and GDT on Occupational Performance and Functional Status in the CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ZEYNEP KOLİT, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CG24
Record Dates: First submitted 2024-01-17; First posted 2024-01-30 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy; Occupational Problems; Cognitive Orientation; Goals
Keywords: cerebral palsy; occupational performance; functional status; CO-OP; goal directed training
MeSH Terms: conditions — Cerebral Palsy; Orientation, Spatial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- coop plus traditional occupational therapy (Experimental): This group received the traditional occupational therapy plus CO-OP approach.
  Interventions: Other: CO-OP; Other: traditional occupational therapy
- GDT plus traditional occupational therapy (Experimental): This group received the traditional occupational therapy plus Goal directed training.
  Interventions: Other: GDT; Other: traditional occupational therapy
- traditional occupational therapy (Other): This group only received the traditional occupational therapy .
  Interventions: Other: traditional occupational therapy

INTERVENTIONS:
Other: CO-OP — With a task-specific and goal-focused CO-OP approach; it is aimed to increase one's skills, to teach to use self-generated cognitive strategies, and to encourage generalization and transfer to new situations and activities.
  Other Names: Cognitive Orientation to Daily Occupational Performance (CO-OP) Approach
  Arms: coop plus traditional occupational therapy
Other: GDT — Goal-directed training included the active implementation of task-specific activities related to the child's functional goals. Focusing on motor learning, GDT is an activity-based approach to therapy that uses meaningful, self-selected goals to provide opportunities for problem solving and indirectly guide the movements necessary to successfully meet task demands
  Other Names: goal directed training
  Arms: GDT plus traditional occupational therapy
Other: traditional occupational therapy — The program included functional one-handed and two-handed training and consisted of advice and treatment aimed at reducing spasticity, improving hand function and activities of daily living, and providing appropriate orthoses. It also includes techniques aimed at improving impairment (e.g., stretching, sensory stimulation) and strengthening activities (e.g., motor training, environmental modification, performing specific target activities) to help participants achieve their individual goals.

SUMMARY:
This study was designed as a three-armed, single-blinded, randomized, controlled trial to examine the effectiveness of CO-OP and GDT interventions on occupational performance and functional status in children with CP compared with their usual care.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of neurological disorders that affect movement, muscle tone, and posture, causing activity limitations that originated in the developing fetal or infant brain that are attributed to non-progressive disorders. Symptoms such as spasticity and contracture in CP cause a decrease in functional skill level with limitations in daily living activities such as learning a new skill or self-dressing and handwriting. In this disease, the simultaneous presence of sensory, cognitive, perceptual, and behavioral impairments significantly undermines the acquisition and execution of functional skills, autonomy in daily living, and active engagement in leisure activities. This study was planned to investigate and compare the impact of CO-OP and GDT on the occupational performance and functional status of children with CP.

ELIGIBILITY:
Inclusion Criteria:

* being between 5-10 years of age
* being diagnosed with CP
* having adequate language abilities to make contact with a therapist and be informed during intervention.

Exclusion Criteria:

* they were receiving any other treatment
* they had been diagnosed with mental retardation
* they had serious vision or hearing problems.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | "up to 12 weeks"
  COPM is used to help individuals describe occupational performance problems and precedence in the areas of self-care, productivity, and leisure, in which they have difficulty performing.
Pediatric Evaluation of Disability Inventory (PEDI): | "up to 12 weeks"
  PEDI is a measurement tool used to evaluate the functional status of children.

CONTACTS AND LOCATIONS:
Overall Officials: zeynep kolit, MSc, Principal Investigator — Hacettepe University; Rüya gül temel, MSc, Principal Investigator — HATAY MUSTAFA KEMAL ÜNİVERSİTESİ; Gamze ekici, PhD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhiye, Turkey (Türkiye)